CLINICAL TRIAL: NCT00800605
Title: Double Blind, Placebo Controlled Phase 3 Study of the Efficacy of an Investigational Vero Cell-Derived Influenza Vaccine to Prevent Culture Confirmed Influenza Infection
Brief Title: Immunogenicity Study of an Inactivated Influenza Vaccine (Split Virus, Vero Cell Derived) to Prevent Culture Confirmed Influenza Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 720802
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Vero cell-derived, trivalent, seasonal influenza vaccine
  Interventions: Biological: Vero cell-derived, trivalent, seasonal influenza vaccine
- 2 (Placebo Comparator): Phosphate-buffered saline
  Interventions: Biological: Placebo: Phosphate-buffered saline

INTERVENTIONS:
Biological: Vero cell-derived, trivalent, seasonal influenza vaccine — Single intramuscular injection
  Arms: 1
Biological: Placebo: Phosphate-buffered saline — Single intramuscular injection
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the efficacy of an investigational Vero cell-derived, trivalent, seasonal influenza vaccine to prevent infection with an influenza virus that is antigenically similar to one of the three strains in the vaccine. Subjects will be randomized in a double-blind fashion to receive a single intramuscular injection of either the investigational vaccine or placebo. Blood will be drawn from all subjects for a determination of hemagglutination inhibition antibody titers on Days 0 and 21, body temperature and injection site reactions will be monitored daily for 7 days. In addition, subjects must return to the clinic promptly to have swab samples of their nose and throat taken whenever they feel flu symptoms and all subjects will be monitored for adverse events until Day 180.

ELIGIBILITY:
Inclusion Criteria:

* Subject has an understanding of the study
* Subject agrees to study provisions
* Subject gives written informed consent prior to study entry
* Subject is accessible by telephone or electronic mail to receive reminders from the study site
* If female and capable of bearing children, subject has a negative urine pregnancy test result within 24 hours of the vaccination on Study Day 0 and agrees to employ adequate birth control measures through the first 60 post-vaccination days.

Exclusion Criteria:

* Subject has any of the risk factors for complications from influenza infection as defined by the Centers for Disease Control and Prevention (CDC, 2008a):

  * Pregnancy
  * Chronic disorders of the pulmonary or cardiovascular system including asthma (hypertension is not considered a high risk condition)
  * Chronic renal disorders
  * Chronic hepatic disorders
  * Chronic hematological disorders
  * Chronic metabolic disorder (including diabetes mellitus and thyroid disorders)
  * Immunosuppression (including immunosuppression caused by medications, congenital etiologies or HIV)
  * Any condition that can compromise respiratory function or the handling of respiratory secretions or that can increase risk for aspiration (e.g., cognitive dysfunction, spinal cord injuries, seizure disorders or other neuromuscular disorders)
  * Residence in nursing home or other chronic care facility that houses persons of any age who have chronic medical conditions
  * Household contact with children aged 0 to 59 months or of someone who is included in the risk categories listed above
  * Employment as a health care worker
* Subject is unable to lead an independent life as a result of either physical or mental handicap
* Subject has a history of severe allergic reactions or anaphylaxis (e.g., urticaria or asthma that is clinically severe)
* Subject has an oral temperature of >= 99.5° F (37.5°C) on the day of vaccination in this study. [NOTE: A subject meeting this exclusion criterion may be rescheduled for vaccination and study entry at a later date provided that certain requirements [in the study protocol] are met)
* Subject has a rash or dermatologic condition or tattoos which may interfere with injection site reaction rating
* Subject has received a blood transfusion, blood products or immunoglobulins within 90 days of study entry
* Subject has received a live vaccine within 4 weeks or inactivated or subunit vaccine within 2 weeks of study entry
* Subject has previously been vaccinated against influenza for the 2008/2009 northern hemisphere influenza season
* Subject has a functional or surgical asplenia
* Subject has a known or suspected problem with alcohol or drug abuse;
* Subject was administered an investigational drug within six weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product
* Subject is a member of the team conducting this study or are in a dependent relationship with the study investigator. Dependent relationships include close relatives (i.e., children, spouse/partner, siblings, parents) as well as employees of the investigator

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7250 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter Bio Science Investigator, MD, Study Director — Baxter Healthcare Corporation
Locations (36):
- United States (36):
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Benchmark Research, Sacramento, California
  - California Research Foundation, San Diego, California
  - Benchmark Research San Francisco, San Francisco, California
  - Radiant Research, Inc, Denver, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Pharmax Research Clinic, Miami, Florida
  - University Clinical Research, Inc, Pembroke Pines, Florida
  - Miami Research Associates, South Miami, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Radiant Research, Inc - Chicago, Chicago, Illinois
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Benchmark Research, Metairie, Louisiana
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Radiant Research, Inc., St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Triangle Medical Research Associates, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Radiant Research - Cincinnati, Cincinnati, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Clinical Research Associates, Inc. - Nashville, Nashville, Tennessee
  - Benchmark Research Austin, Austin, Texas
  - Benchmark Research Ft. Worth, Fort Worth, Texas
  - Benchmark Research San Angeolo, San Angelo, Texas
  - Jean Brown Research / Westside Medical, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - PI-COOR Clinical Research, Burke, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- VCIV: Vero cell-derived, trivalent, seasonal influenza vaccine
  Vero cell-derived, trivalent, seasonal influenza vaccine: Single intramuscular injection
- Placebo: Phosphate-buffered saline
  Placebo: Phosphate-buffered saline: Single intramuscular injection
Period: Overall Study
Arm/Group | VCIV | Placebo
Started | 3626 | 3624
Completed | 3421 | 3415
Not Completed | 205 | 209

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population
Groups:
- Total: Total of all reporting groups
Arm/Group | VCIV | Placebo | Total
Number analyzed (Participants) | 3623 | 3620 | 7243
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (9.7) | 32.1 (9.7) | 32.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1800 | 1755 | 3555
  Male | 1823 | 1865 | 3688
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 616 | 638 | 1254
  Not Hispanic or Latino | 3007 | 2982 | 5989
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 25 | 39
  Asian | 60 | 37 | 97
  Native Hawaiian or Other Pacific Islander | 12 | 10 | 22
  Black or African American | 771 | 741 | 1512
  White | 2746 | 2784 | 5530
  More than one race | 20 | 21 | 41
  Unknown or Not Reported | 0 | 2 | 2
Weight [Mean (Standard Deviation); unit: kg] | 83.6 (22) | 83.3 (21.1) | 83.5 (21.6)
Height [Mean (Standard Deviation); unit: cm] | 171.6 (10) | 171.9 (10.2) | 171.7 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of an Investigational Vero Cell-derived Influenza Vaccine to Prevent Infection With an Influenza Virus That is Antigenically Similar to One of the Three Strains in the Vaccine
Description: The number of subjects developing influenza infection, as confirmed by viral culture and typing of naso-pharyngeal specimens, with a virus that is antigenically similar to one of the strains contained in the vaccine 21 days to 180 days after the date of vaccination.
Time Frame: 180 days
Population: Intent-to-Treat Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3619 | 3617
Participants
  Influenza Infections A/H1N1 Strain | 11 | 52
  Influenza Infections A/H3N2 Strain | 2 | 4
  Influenza Infections B Strains | 0 | 4
  No Influenza Infections | 3606 | 3557

2. Secondary Outcome: Number of Subjects Who Developed Influenza Infection 21 Days to 180 Days Post-vaccination With Infecting Strain Matching the Strains Contained in the Vaccine
Description: Number of subjects with influenza infection confirmed by viral culture and typing and/or RT-PCR analysis of naso-pharyngeal specimens that are antigenically similar to the strains contained in the vaccine
Time Frame: 180 days
Population: Intent-to-Treat Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3619 | 3617
Participants
  Influenza Infection A/H1N1 | 14 | 56
  Influenza Infection A/H3N2 | 2 | 4
  Influenza Infection B | 8 | 20
  No Influenza Infection | 3595 | 3537

3. Secondary Outcome: Number of Subjects Who Developed Influenza Infection Between 21 and 180 Days Post-vaccination, Regardless of Whether the Infecting Strain Matched the Vaccine Strains Antigenically
Description: Number of subjects with influenza infection as confirmed by viral culture and typing of naso-pharyngeal specimens regardless of whether the isolate is antigenically matched to the strains contained in the vaccine
Time Frame: 180 days
Population: Intent-to-Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3619 | 3617
Participants
  Influenza Infection A/H1N1 | 11 | 52
  Influenza Infection A/H3N2 | 2 | 4
  Influenza Infection B | 8 | 18
  No Influenza Infection | 3598 | 3543

4. Secondary Outcome: HIA Titer for Each of the Three Antigens Contained in the Vaccine at Day 21
Time Frame: 21 days
Population: Immunogenicity Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3473 | 3459
Titers
  A/H1N1 | 194.1 [184.4 to 204.3] | 17.7 [17 to 18.4]
  A/H3N2 | 299.7 [285.2 to 314.9] | 22.4 [21.3 to 23.5]
  B | 301.7 [290.5 to 313.4] | 39.3 [37.6 to 41.2]

5. Secondary Outcome: Percentage of Subjects With Seroprotective Antibody Titer [Reciprocal HIA Titer ≥ 40] for Each of the Three Antigens Contained in the Vaccine at Day 21
Time Frame: 21 days
Population: Immunogenicity Analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3473 | 3459
percentage of participants
  A/H1N1 | 88 [86.8 to 89] | 29.8 [28.3 to 31.4]
  A/H3N2 | 93.3 [92.4 to 94.1] | 38.8 [37.2 to 40.5]
  B | 97.1 [96.5 to 97.7] | 56.2 [54.5 to 57.8]

6. Secondary Outcome: Fold Increase of HIA Titer for Each of the Three Antigens Contained in the Vaccine at Day 21 as Compared to Baseline
Time Frame: 21 days
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3473 | 3459
Fold change
  A/H1N1 | 11.11 [10.52 to 11.74] | 1.06 [1.04 to 1.08]
  A/H3N2 | 13.51 [12.85 to 14.2] | 1.01 [1 to 1.02]
  B | 7.58 [7.22 to 7.97] | 1.03 [1.02 to 1.05]

7. Secondary Outcome: Percentage of Subjects Demonstrating Seroconversion to Each of the Three Antigens Contained in the Vaccine at Day 21
Description: Seroconversion is defined as a ≥ 4-fold increase in HIA titer from baseline or a HIA titer ≥ 40 when there is no detectable HIA titer (HIA titer <10) at baseline.
Time Frame: 21 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3473 | 3459
percentage of participants
  A/H1N1 | 70.4 [68.9 to 71.9] | 1.2 [0.9 to 1.6]
  A/H3N2 | 79.1 [77.7 to 80.4] | 0.9 [0.6 to 1.3]
  B | 65.7 [64.1 to 67.3] | 1.3 [1 to 1.7]

8. Secondary Outcome: Frequency and Severity of Occurrence of Any Injection Site Reactions Related to Vaccination
Description: Number of Subjects With Non-Serious Local Reactions During the Entire Follow-Up Period
Time Frame: 180 days
Population: Safety Analysis
Measure: Number; unit: participants
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3623 | 3620
participants
  No Reaction | 1994 | 3309
  Mild | 1354 | 262
  Moderate | 107 | 6
  Severe | 9 | 1
  Unknown | 159 | 42
  Total with Reaction | 1629 | 311

9. Secondary Outcome: Frequency and Severity of Occurrence of Any Injection Site Reactions and Systemic AEs Observed During the Entire 180-day Follow-up Period
Time Frame: 180 days
Population: Safety Analysis
Measure: Number; unit: participants
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3623 | 3620
participants
  Serious AEs | 29 | 27
  Non-Serious Moderate or Severe Systemic AEs | 924 | 858
  Any Non-Serious Systemic AEs | 2176 | 1945
  Non-Serious Moderate or Severe Local AEs | 121 | 7
  Any Non-Serious Local AEs | 1629 | 311

10. Secondary Outcome: Frequency and Severity of Occurrence of Any Systemic Reactions Related to Vaccination
Description: Number of Subjects With Non-Serious Systemic Reactions During the Entire Follow-Up Period
Time Frame: 180 days
Population: Safety Analysis
Measure: Number; unit: participants
Arm/Group | VCIV | Placebo
Number analyzed (Participants) | 3623 | 3620
participants
  No Reaction | 2312 | 2748
  Mild | 957 | 648
  Moderate | 250 | 173
  Severe | 53 | 17
  Unknown | 51 | 34
  Total with Reaction | 1311 | 872

ADVERSE EVENTS:
Arm/Group | VCIV | Placebo
All-Cause Mortality (participants affected / at risk) | 2/3623 | 0/3620
Serious Adverse Events (participants affected / at risk) | 29/3623 | 27/3620
Other Adverse Events (participants affected / at risk) | 2176/3623 | 1945/3620
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VCIV (N=3623) | Placebo (N=3620)
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 4
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Lung injury (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 1 | 0
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pneumonia (Infections and infestations) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Selective abortion (Surgical and medical procedures) | 0 | 3
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Lung injury (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Fallopian tube disorder (Reproductive system and breast disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Uterine enlargement (Reproductive system and breast disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 3 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Chest pain (General disorders) | 1 | 0
Accidental death (General disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VCIV (N=3623) | Placebo (N=3620)
Lymph Node Pain (Blood and lymphatic system disorders) | 3 | 6
Lymphadenopathy (Blood and lymphatic system disorders) | 16 | 28
Ear Discomfort (Ear and labyrinth disorders) | 7 | 5
Ear Pain (Ear and labyrinth disorders) | 41 | 26
Conjunctivitis (Eye disorders) | 6 | 11
Eye Discharge (Eye disorders) | 11 | 3
Eye Irritation (Eye disorders) | 13 | 3
Lacrimation Increased (Eye disorders) | 15 | 15
Ocular Hyperaemia (Eye disorders) | 78 | 38
Abdominal Discomfort (Gastrointestinal disorders) | 14 | 24
Abdominal Pain (Gastrointestinal disorders) | 14 | 11
Abdominal Pain Upper (Gastrointestinal disorders) | 28 | 28
Constipation (Gastrointestinal disorders) | 3 | 8
Diarrhoea (Gastrointestinal disorders) | 114 | 120
Dyspepsia (Gastrointestinal disorders) | 13 | 12
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 212 | 203
Toothache (General disorders) | 15 | 14
Vomiting (Gastrointestinal disorders) | 112 | 105
Chest Discomfort (General disorders) | 11 | 4
Chest Pain (General disorders) | 9 | 12
Chills (General disorders) | 359 | 226
Fatigue (General disorders) | 1189 | 1004
Influenza Like Illness (General disorders) | 36 | 41
Injection Site Erythema (General disorders) | 114 | 27
Injection Site Haematoma (General disorders) | 13 | 11
Injection Site Induration (General disorders) | 125 | 14
Injection Site Pain (General disorders) | 1571 | 274
Injection Site Pruritus (General disorders) | 9 | 1
Injection Site Swelling (General disorders) | 100 | 10
Malaise (General disorders) | 837 | 537
Oedema Peripheral (General disorders) | 2 | 8
Pain (General disorders) | 44 | 40
Pyrexia (General disorders) | 270 | 273
Unevaluable Event (General disorders) | 6 | 7
Seasonal Allergy (Infections and infestations) | 11 | 11
Bronchitis (Infections and infestations) | 23 | 29
Ear Infection (Infections and infestations) | 6 | 8
Gastroenteritis (Infections and infestations) | 18 | 25
Influenza (Infections and infestations) | 3 | 6
Laryngitis (Infections and infestations) | 10 | 5
Nasopharyngitis (Infections and infestations) | 67 | 66
Oral Herpes (Immune system disorders) | 5 | 11
Otitis Media (Infections and infestations) | 10 | 4
Pharyngitis (Infections and infestations) | 18 | 21
Pharyngitis Streptococcal (Infections and infestations) | 13 | 19
Pneumonia (Infections and infestations) | 8 | 1
Rhinitis (Infections and infestations) | 19 | 23
Sinusitis (Infections and infestations) | 52 | 46
Tonsillitis (Infections and infestations) | 3 | 6
Tooth Abscess (Infections and infestations) | 10 | 2
Tooth Infection (Infections and infestations) | 8 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 105 | 118
Urinary Tract Infection (Infections and infestations) | 13 | 19
Viral Infection (Infections and infestations) | 18 | 26
Viral Upper Respiratory Tract Infection (Infections and infestations) | 25 | 29
Contusion (Injury, poisoning and procedural complications) | 6 | 6
Joint Sprain (Injury, poisoning and procedural complications) | 6 | 10
Limb Injury (Injury, poisoning and procedural complications) | 6 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 9 | 8
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 9 | 6
Procedural Pain (Injury, poisoning and procedural complications) | 16 | 14
Skin Laceration (Injury, poisoning and procedural complications) | 11 | 7
Blood Pressure Increased (Investigations) | 54 | 55
Body Temperature Increased (Investigations) | 21 | 29
Anorexia (Metabolism and nutrition disorders) | 10 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 335 | 217
Back Pain (Musculoskeletal and connective tissue disorders) | 42 | 48
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 15 | 11
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 10 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 1042 | 648
Neck Pain (Musculoskeletal and connective tissue disorders) | 18 | 18
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 19 | 16
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 3 | 6
Dizziness (Nervous system disorders) | 31 | 42
Headache (Nervous system disorders) | 1408 | 1292
Migraine (Nervous system disorders) | 16 | 8
Paraesthesia (Nervous system disorders) | 3 | 6
Sinus Headache (Nervous system disorders) | 42 | 32
Anxiety (Psychiatric disorders) | 11 | 9
Depression (Psychiatric disorders) | 14 | 11
Insomnia (Psychiatric disorders) | 21 | 16
Dysmenorrhoea (Reproductive system and breast disorders) | 17 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 470 | 476
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 15
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 236 | 243
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 529 | 506
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 10 | 15
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 8 | 24
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 22 | 17
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 17
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 75 | 57
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 175 | 175
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 52 | 67
Sneezing (Respiratory, thoracic and mediastinal disorders) | 57 | 69
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 34 | 23
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 3 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 265 | 198
Night Sweats (Skin and subcutaneous tissue disorders) | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes